CLINICAL TRIAL: NCT00939978
Title: Effect of Preoperative Recombinant Human Erythropoietin on Transfusion Risk in Valvular Heart Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Young-Lan Kwak/Professor, Severance Hospital
Other Study IDs: 4-2008-0427
Record Dates: First submitted 2009-07-14; First posted 2009-07-15 (Estimated); Last update posted 2010-10-07 (Estimated); Status verified 2010-10

CONDITIONS: Cardiac Surgery

ARMS (2):
- Venoferrum (Active Comparator)
  Interventions: Drug: rhEPO
- saline (Placebo Comparator)
  Interventions: Drug: rhEPO

INTERVENTIONS:
Drug: rhEPO — recombinant human erythropoietin(rhEPO)

SUMMARY:
The administration of rhEPO on the one day before cardiac surgery will be effective to decrease the bleeding due to the surgery.

ELIGIBILITY:
Inclusion Criteria:

* The 90 patients who are planned to have the heart surgery during this study period.(minimum age 20)

Exclusion Criteria:

* Uncontrolled hypertension(diastolic blood pressure(DBP)>100 mmHg), Hct > 45%, Plt. count)>450,000
* There are no history of seizure, thrombus, cancer, acute hepatitis, alcoholism, peripheral blood vessel disease, pure red blood cell dysfunction, liver function failure, chronic multiple arthritis.
* No pregnancy, acute hyper parathyroidism.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2009-04; Primary Completion 2010-06 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Severance hospital, Seoul, South Korea